CLINICAL TRIAL: NCT00033397
Title: Contrast-Enhanced Breast MRI, MRS, And Correlative Science Studies To Characterize Tumor Response In Patients Undergoing Neoadjuvant Treatment For Locally Advanced Breast Cancer
Brief Title: Diagnostic Procedures in Women With Locally Advanced Breast Cancer Who Are Receiving Chemotherapy Before Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150007; CALGB-150007; CDR0000069280 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Biopsy; Magnetic Resonance Spectroscopy; High-Energy Shock Waves; Gadolinium DTPA; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm A: Patients receive an injection of gadopentetate dimeglumine and undergo magnetic resonance imaging (MRI) of the breast before initiation, 1-3 days after initiation, and then after completion of neoadjuvant anthracycline-based chemotherapy and prior to surgery. Patients who previously received a taxane also undergo an additional contrast-enhanced MRI scan.
  Mammograms and possibly ultrasounds are performed prior to and after chemotherapy (before surgery).
  Patients are followed every 6 months for 5 years and then annually for up to 10 years.
  Interventions: Procedure: biopsy; Procedure: magnetic resonance imaging; Procedure: radiomammography; Procedure: ultrasound imaging; Radiation: gadopentetate dimeglumine; Drug: chemotherapy

INTERVENTIONS:
Procedure: biopsy
Procedure: magnetic resonance imaging
Procedure: radiomammography
Procedure: ultrasound imaging
Radiation: gadopentetate dimeglumine
Drug: chemotherapy

SUMMARY:
RATIONALE: Comparing results of diagnostic procedures performed before, during, and after chemotherapy may help doctors predict a patient's response to treatment and help plan the most effective treatment.

PURPOSE: Diagnostic trial to study magnetic resonance imaging (MRI) and biomarkers in women who are receiving chemotherapy before surgery for locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Support accrual to the ACRIN-6657/CALGB-150012 magnetic resonance imaging (MRI) correlative science study.
* Determine whether molecular markers, alone or in combination with MRI, at the time of diagnosis or early in the course of therapy, predict 3-year disease-free survival (DFS) in women with locally advanced breast cancer who are receiving neoadjuvant chemotherapy.
* Identify two groups of participants who have statistically different 3-year DFS, based on 1 or more biomarkers, including MRI.
* Determine whether biomarkers, in combination with MRI, early in the course of chemotherapy, improve the prediction of 3-year DFS and are at least as good of a predictor of DFS as residual disease at the time of surgery in these patients.
* Determine whether molecular markers are associated with specific imaging patterns seen on MRI of these patients.
* Predict response with MRI results and marker data from cell cycle check points, proliferation, angiogenesis, hormone receptors, and molecular profiles in these patients.

Secondary

* Determine the molecular predictors of lack of radiologic complete response (CR) in HER-2/neu negative patients (immunohistochemistry [IHC] score of 0, 1+, 2 and fluorescence in situ hybridization [FISH] not amplified) after a neoadjuvant anthracycline-based regimen.
* Determine the molecular predictors of lack of radiologic CR in HER-2/neu positive patients (IHC 3+ or FISH amplified > 2.0) after a neoadjuvant anthracycline-based regime followed by a taxane alone regimen or in combination with trastuzumab.
* Determine the molecular predictors of complete magnetic resonance imaging radiologic response to a neoadjuvant anthracycline-based regimen when gene expression profiling is performed in a sequential, real-time fashion.

OUTLINE: This is a diagnostic, multicenter study conducted concurrently with CALGB-150012/ACRIN-6657 imaging protocol and concurrently with neoadjuvant anthracycline-based chemotherapy.

Patients receive an injection of gadopentetate dimeglumine and undergo magnetic resonance imaging (MRI) of the breast before initiation, 1-3 days after initiation, and then after completion of neoadjuvant anthracycline-based chemotherapy and prior to surgery. Patients who previously received a taxane also undergo an additional contrast-enhanced MRI scan.

Patients undergo biopsies before initiation and at the time of surgery. Patients also undergo blood draws at the time of the first biopsy and prior to surgery. Serum and tissue samples are used to assess biomarkers of genetic instability, cell cycle progression and cellular proliferation as predictors for anthracycline responsiveness, markers of apoptotic potential as predictors for taxane responsiveness in vivo, angiogenesis, hormone receptors, and molecular profiles using immunohistochemical methods.

Mammograms and possibly ultrasounds are performed prior to and after chemotherapy (before surgery).

Patients are followed every 6 months for 5 years and then annually for up to 10 years.

PROJECTED ACCRUAL: A total of 384 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed adenocarcinoma of the breast by core needle biopsy, incisional biopsy, or fine needle aspiration (FNA)

  * Incisional biopsy must result in < 10% removal of gross residual disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan OR
* Nonmeasurable disease
* Meets one of the following staging criteria:

  * Stage II or III disease
  * T4, any N, M0, including clinical or pathologic inflammatory disease
  * Regional stage IV disease where supraclavicular/infraclavicular lymph nodes are only site of metastasis
* No clinical or imaging evidence of distant metastasis
* Metaplastic carcinomas allowed
* Synchronous bilateral primaries allowed if the more advanced tumor meets staging criteria
* Patients for whom FNA was used to confirm initial diagnosis must have histologically confirmed invasive carcinoma by the start of chemotherapy
* Her-2/neu status known
* Currently receiving neoadjuvant chemotherapy consisting of a taxane-based regimen alone or followed by an anthracycline-based regimen
* Concurrent enrollment in the ACRIN-6657/CALGB-150012 imaging protocol required
* Hormone receptor status:

  * Any estrogen receptor or progesterone receptor status

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female Cardiovascular
* No uncontrolled or severe cardiovascular disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* No ferromagnetic prostheses including the following:

  * Metallic implants not compatible with a magnetic resonance imaging machine
  * Heart valves
  * Aneurysm clips
  * Orthopedic prosthesis
  * Any metallic fragments anywhere in the body

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy to the ipsilateral breast for this malignancy

Endocrine therapy

* At least 4 weeks since prior tamoxifen or raloxifene

Radiotherapy

* No prior radiotherapy to the ipsilateral breast for this malignancy

Other

* No other prior cytotoxic regimens

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2002-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05-01 (Actual)

PRIMARY OUTCOMES:
response | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura J. Esserman, MD, MBA, Study Chair — University of California, San Francisco
Locations (5):
- United States (5):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Background] Carey LA, Oh D, Sawyer L, et al.: Gene expression subtype and p53 mutational status are correlated among neoadjuvantly treated breast cancers in UNC LCCC9819 and I-SPY1 (CALGB 150007/ACRIN 6657). [Abstract] J Clin Oncol 24 (Suppl 18): A-10048, 552s, 2006.
- [Result] Esserman LJ, Berry DA, Cheang MC, Yau C, Perou CM, Carey L, DeMichele A, Gray JW, Conway-Dorsey K, Lenburg ME, Buxton MB, Davis SE, van't Veer LJ, Hudis C, Chin K, Wolf D, Krontiras H, Montgomery L, Tripathy D, Lehman C, Liu MC, Olopade OI, Rugo HS, Carpenter JT, Livasy C, Dressler L, Chhieng D, Singh B, Mies C, Rabban J, Chen YY, Giri D, Au A, Hylton N; I-SPY 1 TRIAL Investigators. Chemotherapy response and recurrence-free survival in neoadjuvant breast cancer depends on biomarker profiles: results from the I-SPY 1 TRIAL (CALGB 150007/150012; ACRIN 6657). Breast Cancer Res Treat. 2012 Apr;132(3):1049-62. doi: 10.1007/s10549-011-1895-2. Epub 2011 Dec 25. PMID 22198468
- [Result] Esserman LJ, Berry DA, DeMichele A, Carey L, Davis SE, Buxton M, Hudis C, Gray JW, Perou C, Yau C, Livasy C, Krontiras H, Montgomery L, Tripathy D, Lehman C, Liu MC, Olopade OI, Rugo HS, Carpenter JT, Dressler L, Chhieng D, Singh B, Mies C, Rabban J, Chen YY, Giri D, van 't Veer L, Hylton N. Pathologic complete response predicts recurrence-free survival more effectively by cancer subset: results from the I-SPY 1 TRIAL--CALGB 150007/150012, ACRIN 6657. J Clin Oncol. 2012 Sep 10;30(26):3242-9. doi: 10.1200/JCO.2011.39.2779. Epub 2012 May 29. PMID 22649152
- [Result] Lin C, Buxton MB, Moore D, Krontiras H, Carey L, DeMichele A, Montgomery L, Tripathy D, Lehman C, Liu M, Olapade O, Yau C, Berry D, Esserman LJ; I-SPY TRIAL Investigators. Locally advanced breast cancers are more likely to present as Interval Cancers: results from the I-SPY 1 TRIAL (CALGB 150007/150012, ACRIN 6657, InterSPORE Trial). Breast Cancer Res Treat. 2012 Apr;132(3):871-9. doi: 10.1007/s10549-011-1670-4. Epub 2011 Jul 28. PMID 21796368
- [Result] Esserman LJ, Perou C, Cheang M, et al.: Breast cancer molecular profiles and tumor response of neoadjuvant doxorubicin and paclitaxel: The I-SPY TRIAL (CALGB 150007/150012, ACRIN 6657). [Abstract] J Clin Oncol 27 (Suppl 15): A-LBA515, 2009.
- [Result] Hylton N, Blume J, Gatsonis C, et al.: MRI tumor volume for predicting response to neoadjuvant chemotherapy in locally advanced breast cancer: findings from ACRIN 6657/CALGB 150007. [Abstract] J Clin Oncol 27 (Suppl 15): A-529, 2009.
- [Result] Lin C, Moore D, DeMichele A, et al.: Detection of locally advanced breast cancer in the I-SPY TRIAL (CALGB 150007/150012, ACRIN 6657) in the interval between routine screening. [Abstract] J Clin Oncol 27 (Suppl 15): A-1503, 2009.
- [Result] Pradhan SM, Carey L, Edmiston S, et al.: P53 mutation and differential response to neoadjuvant chemotherapy in women with locally advanced breast cancer: results from the I-SPY trial (CALGB 150007/1500012 and ACRIN 6657). [Abstract] J Clin Oncol 27 (Suppl 15): A-11099, 2009.
- [Result] Van 't Veer LJ, Das D, DeMichele A, et al.: Neoadjuvant response in the context of a biologically defined low or high risk tumor has a different clinical consequence, the I-SPY trial (CALGB 150007/150012, ACRIN 6657). [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-2003, 2009.
- [Result] Wolf DM, Das D, Lenburg ME, et al.: From the lab to the clinic: gene-expression profiles that are associated with Mek-inhibitor sensitivity in vitro are coordinately co-expressed in breast cancer biopsy samples from the I-SPY Trial (CALGB 150007/150012, ACRIN 6657). [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-2042, 2009.
- [Result] Esserman LJ, van't Veer LJ, Perou C, et al.: Biology of breast cancers that present as interval cancers and at young age should inform how we approach early detection and prevention. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-6034, 2008.
- [Result] Gomez RE, Zakhireh J, Moore D, et al.: Sentinel node biopsy performed in the neoadjuvant setting for breast cancer: results from the I-SPY TRIAL (CALGB 150007/150012 & ACRIN 6657). [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-202, 2008.
- [Result] Livasy C, Carey L, DeMichele A, et al.: Influence of anthracycline- and taxane-based neoadjuvant chemotherapy on tumor HER2 protein expression in locally advanced breast cancers: results from the I-SPY TRIAL (CALGB 150007/150012 & ACRIN 6657). [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-703, 2008.
- [Result] Livasy C, Carey L, DeMichele A, et al.: Biomarkers associated with pathologic complete response to neoadjuvant chemotherapy in women with locally advanced breast cancer: results from the I-SPY TRIAL (CALGB 150007/150012 & ACRIN 6657). [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-5102, 2008.
- [Result] Conway K, Edmiston SN, Tolbert D, et al.: Preliminary evaluation of p53 mutation type, tumor characteristics and clinical response among neoadjuvantly treated breast cancer patients in I-SPY1 (CALGB 150007/ACRIN 6657). [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-3029, S134, 2006.
- [Derived] Magbanua MJ, Wolf DM, Yau C, Davis SE, Crothers J, Au A, Haqq CM, Livasy C, Rugo HS; I-SPY 1 TRIAL Investigators; Esserman L, Park JW, van 't Veer LJ. Serial expression analysis of breast tumors during neoadjuvant chemotherapy reveals changes in cell cycle and immune pathways associated with recurrence and response. Breast Cancer Res. 2015 May 29;17(1):73. doi: 10.1186/s13058-015-0582-3. PMID 26021444